CLINICAL TRIAL: NCT04014400
Title: A Randomized Controlled Trial Comparing Suprathel Versus Xeroform for the Management of Pediatric and Adult Split Thickness Skin Graft Donor Sites
Brief Title: Suprathel Versus Xeroform for the Management of Skin Graft Donor Sites
Acronym: Suprathel
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We observed that using the Suprathel dressing required additional treatment of the wound and had a longer healing time than the standard of care Xeroform dressing; it did not dry the wound out properly to promote healing.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-1048
Record Dates: First submitted 2019-07-01; First posted 2019-07-10 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Burns; Skin Graft Complications; Skin; Deformity
Keywords: skin graft; suprathel; xeroform; burn; donor site
MeSH Terms: conditions — Burns; Skin Abnormalities | interventions — poly(lactide-co-trimethylenecarbonate-co-epsilon-caprolactone)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprathel (Experimental): Once hemostasis is obtained, the Suprathel material will be handled with a new pair of sterile gloves. It will be cut so that the material extends 1-2 cm beyond the donor site margins, then applied to the donor site. The Suprathel will be secured with a protective layer of Rylon extending 1-2 cms beyond the margins of the Suprathel. The primary dressing will be covered with cotton gauze (4x4 fluff gauze pads) and wrapped with rolled gauze). The outer dressing will be changed 7-10 days post-op. The Suprathel and Rylon will remain in place until they can be easily peeled off. To facilitate the pain-free and easy removal of the primary Suprathel dressing, practioners will apply Vaseline or lotion to saturate and loosen the material. The patients will be followed on average about once per week in an outpatient clinic until the Suprathel (and Rylon) are removed, but they may continue to be seen until the STSG is fully healed.
  Interventions: Other: Suprathel or Xeroform donor site application
- Xeroform (Active Comparator): After hemostasis occurs, the Xeroform dressing will be handled with a new pair of sterile gloves and cut so that the material extends 1-2 cm beyond the donor site margins, then applied to the donor site. The primary dressing will be covered with cotton gauze (4x4 fluff gauze pads) and wrapped with rolled gauze (Kerlix). The outer dressing will be changed 7-10 days post-op. The Xeroform will remain in place until it can be easily peeled off. To facilitate the pain-free and easy removal of the Xeroform dressing, practioners may apply Vaseline or lotion to saturate and loosen the material. The patients will be followed on average about once per week in an outpatient clinic until the Xeroform is removed, but they may continue to be seen until the STSG is fully healed.
  Interventions: Other: Suprathel or Xeroform donor site application

INTERVENTIONS:
Other: Suprathel or Xeroform donor site application — The surgical procedure for recovery of a skin graft will be the same for all patients as follows. Once the patient is taken to the operating room, the selected donor site will be prepared and harvested with a Zimmer Dermatome set at 0.007 to 0.009 thousands of an inch for pediatric patients and 0.12 to 0.14 thousands for adult patients. After the harvesting procedure, the donor site will be covered with Telfa saturated with 1:10,000 epinephrine in normal saline until hemostasis is achieved. The Telfa will be irrigated off the donor site with the epinephrine saline solution. The surgeon will don a new pair of sterile gloves to handle the donor site dressing. The randomized dressing will be applied over the hemostatic donor site with an approximate 1-2cm border. Next, the wound will be dressed with 4x4 cotton gauze pads (fluffs), rolled gauze (Kerlix) and either Coban or BandNet.

SUMMARY:
The investigators aim to study whether Suprathel, a synthetic temporary skin substitute developed by PolyMedics Innovations GmBH aids in the management of patient pain and wound healing when compared to the current standard dressing used of a primary Xeroform dressing.

DETAILED DESCRIPTION:
Acute burn and donor site dressing changes are among the most traumatic and painful procedures performed on awake children and adults (7, 8). As a result, it is important to utilize dressings that: 1) stabilize open burn wounds and donor sites; 2) limit the frequency of dressing changes; 3) optimize burn wound and donor site healing; and 4) minimize scarring. Anecdotal evidence and a growing body of literature suggest that Suprathel may offer superior pain control and a decreased frequency of dressing changes, when compared to Xeroform.

At Children's Hospital Colorado, the standard of care is to use Xeroform to dress split thickness skin grafts and donor sites. Xeroform is an inexpensive, bacteriostatic, non-adherent petroleum gauze dressing that is supplied in strips, sheets and rolls. It is used to protect freshly skin grafted areas and donor sites, it is then covered with gauze followed by BandNet. When Xeroform is applied to a split thickness donor site, it adheres to the open wound bed, where it is allowed to dry out. As the donor site heals, the Xeroform begins to separate from the wound bed, until the Xeroform eventually sloughs off.

Suprathel is a biosynthetic dressing developed by PolyMedics Innovations in Germany. Potential advantages to the use of Suprathel include its water solubility, elongation capacity, and porosity, which prevents fluid accumulation at the burn site. In a prior study, Suprathel was associated with favorable burn scar formation (improved Vancouver Scar Scale Scores) and decreased pain with dressing changes. In another study, adolescent and adult burn patients dressed in Suprathel reported significantly less pain than those who were dressed in Mepilex dressings. In post-treatment surveys, patients preferred the use of Suprathel when compared to Mepitel. In a study that compared Suprathel to other standard burn dressings, there was no statistical difference in wound healing, scar formation, and epithelization. Given the limitations in sample size and scarce pediatric data in prior studies, further research is necessary to determine the efficacy of Suprathel in the pediatric population and whether this is a dressing material that should be offered to hospital patients.

New outpatients and inpatients who meet study inclusion criteria and require split-thickness skin grafting, will be randomized into the Suprathel group or the control group on the day of surgery. The investigators will use even calendar operative days for Suprathel and odd calendar operative days for Xeroform. Parental consent and/or patient assent will be obtained prior to the operative procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children 31 days old -17 years old
* Have a burn injury or open wound of any percentage TBSA
* Require a skin graft

Exclusion Criteria:

* allergy to one of the dressings involved in the study,
* burn in close proximity to the donor site,
* the donor site has been harvested in a previous surgery,
* prisoners,
* children under the protection of the department of human services,
* pregnant women,
* those with impaired decision-making capacity.

Ages: 31 Days to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Change in Pain as Assessed by Bieri Faces Scale | Weekly change in pain for 12 weeks
  The Bieri faces scale was developed in 1990 for children to self-report their pain levels by selecting a face corresponding to their pain severity. The Bieri faces scale has been validated in children >5 years old. Children are asked to select one of 7 faces ranging from no pain to worst possible pain.
Pain Before Dressing Change as assessed by r-FLACC | Weekly change in pain for 12 weeks
  Burn clinic providers will rate each child's pain before and after dressing changes using the r-FLACC scoring tool. Scores range from 0-2, with higher scores indicating more pain.
Pain After Dressing Change as assessed by r-FLACC | Weekly change in pain for 12 weeks
  Burn clinic providers will rate each child's pain before and after dressing changes using the r-FLACC scoring tool. Scores range from 0-2, with higher scores indicating more pain.
POSAS Scale Score | Weekly change in scar from 3rd week to 12 weeks
  This scale is a validated tool that will be adapted so that parents and providers score the child's wound based on several criteria. The observer/provider will evaluate vascularization, pigmentation, thickness, surface roughness, pliability, and surface area. The patient's parents will score six items: pain, pruritus, color, thickness, relief, and pliability. It is widely used in the burn literature to evaluate and report on the appearance of healed burn scars. Moreover, it routinely used in the burn clinic at CHCO to assess and serially document changes in the appearance of burn scars over time.
Change in Pain as Assessed using Visual Analog Scale | Weekly change in pain for 12 weeks
  The visual analog scale is widely used to assess pain in the burn population. It was developed by Huskisson in 1974 and evaluates pain on a scale of 0 to 10; it has been validated in children >7 years old.
PROMIS Pain Interference Survey | Weekly change in pain interference for 12 weeks
  The PROMIS pain interference survey (short form) is an eight-question survey developed by the NIH to assess pain control over the past week in children >8 years old.
PROMIS Pain Interference Proxy Survey | Weekly change in pain interference for 12 weeks
  The PROMIS pain interference proxy form (short form) is an eight-question survey developed by the NIH to assess parents' perceptions of their child's pain control over the past week.
Pain Diary application (PainScale) | Day 1 through Day 7-10 Post-op
  This is a free, downloadable application for androids and iPhones. It will be used by patients and/or their parents to document their pain severity, location, and medication use. Each report will be sent to the study coordinator via a HIPAA compliant server. Parents or patients will be asked to document their pain levels and pain medication use postoperatively for the first 7-10 days (until their first clinic appointment).

SECONDARY OUTCOMES:
Infection | 1 day (study visit) per week up to 12 weeks
  Presence of absence of infection at the donor site (s) based on odor, rash, deep red appearance or pruritus--these wounds will typically not be cultured.
Cost of dressings | 12 weeks
  Overall dressing cost
Heal time | 12 weeks
  number of clinic visits until the burn provider or plastics PA considers the donor site(s) healed
re-epithelialization | 12 weeks
  Number of days to re-epithelialization
Burn Itch Severity as assessed by Itch Man Scale | 12 weeks
  The Itch man scale is validated in patients 6 years or older and uses a Likert scale to quantify the degree of itchiness. A score of 0 is not itchy at all, a score of 4 reflects the most itchy.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Moulton, MD, Principal Investigator — Children's Hospital Colorado
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reed JL, Pomerantz WJ. Emergency management of pediatric burns. Pediatr Emerg Care. 2005 Feb;21(2):118-29. doi: 10.1097/01.pec.0000159058.95424.0d. No abstract available. PMID 15699824
- [Background] Hundeshagen G, Collins VN, Wurzer P, Sherman W, Voigt CD, Cambiaso-Daniel J, Nunez Lopez O, Sheaffer J, Herndon DN, Finnerty CC, Branski LK. A Prospective, Randomized, Controlled Trial Comparing the Outpatient Treatment of Pediatric and Adult Partial-Thickness Burns with Suprathel or Mepilex Ag. J Burn Care Res. 2018 Feb 20;39(2):261-267. doi: 10.1097/BCR.0000000000000584. PMID 28557869
- [Background] Rashaan ZM, Krijnen P, Allema JH, Vloemans AF, Schipper IB, Breederveld RS. Usability and effectiveness of Suprathel(R) in partial thickness burns in children. Eur J Trauma Emerg Surg. 2017 Aug;43(4):549-556. doi: 10.1007/s00068-016-0708-z. Epub 2016 Jul 18. PMID 27432172
- [Background] Kaartinen IS, Kuokkanen HO. Suprathel((R)) causes less bleeding and scarring than Mepilex((R)) Transfer in the treatment of donor sites of split-thickness skin grafts. J Plast Surg Hand Surg. 2011 Sep;45(4-5):200-3. doi: 10.3109/2000656X.2011.583515. PMID 22150140
- [Background] Everett M, Massand S, Davis W, Burkey B, Glat PM. Use of a copolymer dressing on superficial and partial-thickness burns in a paediatric population. J Wound Care. 2015 Jul;24(7):S4-8. doi: 10.12968/jowc.2015.24.Sup7.S4. PMID 26198721
- [Background] Hansbrough W, Dore C, Hansbrough JF. Management of skin-grafted burn wounds with Xeroform and layers of dry coarse-mesh gauze dressing results in excellent graft take and minimal nursing time. J Burn Care Rehabil. 1995 Sep-Oct;16(5):531-4. doi: 10.1097/00004630-199509000-00012. PMID 8537426
- [Background] Gee Kee E, Kimble RM, Cuttle L, Stockton K. Comparison of three different dressings for partial thickness burns in children: study protocol for a randomised controlled trial. Trials. 2013 Nov 25;14:403. doi: 10.1186/1745-6215-14-403. PMID 24274190
- [Background] Piatkowski A, Drummer N, Andriessen A, Ulrich D, Pallua N. Randomized controlled single center study comparing a polyhexanide containing bio-cellulose dressing with silver sulfadiazine cream in partial-thickness dermal burns. Burns. 2011 Aug;37(5):800-4. doi: 10.1016/j.burns.2011.01.027. Epub 2011 Feb 23. PMID 21349646
- [Background] Vloemans AF, Hermans MH, van der Wal MB, Liebregts J, Middelkoop E. Optimal treatment of partial thickness burns in children: a systematic review. Burns. 2014 Mar;40(2):177-90. doi: 10.1016/j.burns.2013.09.016. Epub 2013 Nov 26. PMID 24290852
- [Background] Markl P, Prantl L, Schreml S, Babilas P, Landthaler M, Schwarze H. Management of split-thickness donor sites with synthetic wound dressings: results of a comparative clinical study. Ann Plast Surg. 2010 Nov;65(5):490-6. doi: 10.1097/SAP.0b013e3181d37624. PMID 20841998
- [Background] Cunningham NR, Kashikar-Zuck S, Mara C, Goldschneider KR, Revicki DA, Dampier C, Sherry DD, Crosby L, Carle A, Cook KF, Morgan EM. Development and validation of the self-reported PROMIS pediatric pain behavior item bank and short form scale. Pain. 2017 Jul;158(7):1323-1331. doi: 10.1097/j.pain.0000000000000914. PMID 28394851
- [Background] Liu Y, Yuan C, Wang J, Brown JG, Zhou F, Zhao X, Shen M, Hinds PS. Comparability of the Patient-Reported Outcomes Measurement Information System Pediatric short form symptom measures across culture: examination between Chinese and American children with cancer. Qual Life Res. 2016 Oct;25(10):2523-2533. doi: 10.1007/s11136-016-1312-8. Epub 2016 May 10. PMID 27165148
- [Background] Brandon TG, Becker BD, Bevans KB, Weiss PF. Patient-Reported Outcomes Measurement Information System Tools for Collecting Patient-Reported Outcomes in Children With Juvenile Arthritis. Arthritis Care Res (Hoboken). 2017 Mar;69(3):393-402. doi: 10.1002/acr.22937. PMID 27159889
- [Background] Bieri D, Reeve RA, Champion DG, Addicoat L, Ziegler JB. The Faces Pain Scale for the self-assessment of the severity of pain experienced by children: development, initial validation, and preliminary investigation for ratio scale properties. Pain. 1990 May;41(2):139-150. doi: 10.1016/0304-3959(90)90018-9. PMID 2367140
- [Background] Baxt C, Kassam-Adams N, Nance ML, Vivarelli-O'neill C, Winston FK. Assessment of pain after injury in the pediatric patient: child and parent perceptions. J Pediatr Surg. 2004 Jun;39(6):979-83; discussion 979-83. doi: 10.1016/j.jpedsurg.2004.02.031. PMID 15185239
- [Background] Cummings EA, Reid GJ, Finley AG, McGrath PJ, Ritchie JA. Prevalence and source of pain in pediatric inpatients. Pain. 1996 Nov;68(1):25-31. doi: 10.1016/S0304-3959(96)03163-6. PMID 9251995
- [Background] Busche MN, Thraen AJ, Gohritz A, Rennekampff HO, Vogt PM. Burn Scar Evaluation Using the Cutometer(R) MPA 580 in Comparison to "Patient and Observer Scar Assessment Scale" and "Vancouver Scar Scale". J Burn Care Res. 2018 Jun 13;39(4):516-526. doi: 10.1093/jbcr/irx009. PMID 29596600
- [Background] Highton L, Wallace C, Shah M. Use of Suprathel(R) for partial thickness burns in children. Burns. 2013 Feb;39(1):136-41. doi: 10.1016/j.burns.2012.05.005. Epub 2012 Jun 13. PMID 22698841
- [Background] Monstrey S, Hoeksema H, Verbelen J, Pirayesh A, Blondeel P. Assessment of burn depth and burn wound healing potential. Burns. 2008 Sep;34(6):761-9. doi: 10.1016/j.burns.2008.01.009. Epub 2008 Jun 3. PMID 18511202
- [Background] Voepel-Lewis T, Malviya S, Tait AR, Merkel S, Foster R, Krane EJ, Davis PJ. A comparison of the clinical utility of pain assessment tools for children with cognitive impairment. Anesth Analg. 2008 Jan;106(1):72-8, table of contents. doi: 10.1213/01.ane.0000287680.21212.d0. PMID 18165556
- [Background] van der Wal MB, Tuinebreijer WE, Bloemen MC, Verhaegen PD, Middelkoop E, van Zuijlen PP. Rasch analysis of the Patient and Observer Scar Assessment Scale (POSAS) in burn scars. Qual Life Res. 2012 Feb;21(1):13-23. doi: 10.1007/s11136-011-9924-5. Epub 2011 May 20. PMID 21598065
- [Background] Schwarze H, Kuntscher M, Uhlig C, Hierlemann H, Prantl L, Ottomann C, Hartmann B. Suprathel, a new skin substitute, in the management of partial-thickness burn wounds: results of a clinical study. Ann Plast Surg. 2008 Feb;60(2):181-5. doi: 10.1097/SAP.0b013e318056bbf6. PMID 18216512
- [Background] Beltramini A, Milojevic K, Pateron D. Pain Assessment in Newborns, Infants, and Children. Pediatr Ann. 2017 Oct 1;46(10):e387-e395. doi: 10.3928/19382359-20170921-03. PMID 29019634
- [Background] Morris V, Murphy LM, Rosenberg M, Rosenberg L, Holzer CE 3rd, Meyer WJ 3rd. Itch assessment scale for the pediatric burn survivor. J Burn Care Res. 2012 May-Jun;33(3):419-24. doi: 10.1097/BCR.0b013e3182372bfa. PMID 22561307